CLINICAL TRIAL: NCT05862818
Title: Can Food Timing Reduce Your Diabetes Risk?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023P001063
Record Dates: First submitted 2023-04-17; First posted 2023-05-17 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Dietary Habits
Keywords: Glucose tolerance; Diet-induced thermogenesis; Fat tolerance
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Day shift protocol with diet A (Experimental): Day shift protocol with diet A condition. Since this is a single-blind study, the details of the meal conditions cannot be released during the recruitment stage but will be made public once enrollment closes.
  Interventions: Behavioral: Day shift protocol - Diet order A-B; Behavioral: Day shift protocol - Diet order B-A
- Day shift protocol with diet B (Experimental): Day shift protocol with diet B condition. Since this is a single-blind study, the details of the meal conditions cannot be released during the recruitment stage but will be made public once enrollment closes.
  Interventions: Behavioral: Day shift protocol - Diet order A-B; Behavioral: Day shift protocol - Diet order B-A
- Night shift protocol with diet A (Experimental): Night shift protocol with diet A condition. Since this is a single-blind study, the details of the meal conditions cannot be released during the recruitment stage but will be made public once enrollment closes.
  Interventions: Behavioral: Night shift protocol - Diet order A-B; Behavioral: Night shift protocol - Diet order B-A
- Night shift protocol with diet B (Experimental): Night shift protocol with diet B condition. Since this is a single-blind study, the details of the meal conditions cannot be released during the recruitment stage but will be made public once enrollment closes.
  Interventions: Behavioral: Night shift protocol - Diet order A-B; Behavioral: Night shift protocol - Diet order B-A

INTERVENTIONS:
Behavioral: Day shift protocol - Diet order A-B — Research participants will be assigned to day shift condition and Diet A-B order condition.
  Arms: Day shift protocol with diet A; Day shift protocol with diet B
Behavioral: Day shift protocol - Diet order B-A — Research participants will be assigned to day shift condition and Diet B-A order condition.
  Arms: Day shift protocol with diet A; Day shift protocol with diet B
Behavioral: Night shift protocol - Diet order A-B — Research participants will be assigned to simulated night shift condition and Diet A-B order condition.
  Arms: Night shift protocol with diet A; Night shift protocol with diet B
Behavioral: Night shift protocol - Diet order B-A — Research participants will be assigned to simulated night shift condition and Diet B-A order condition.
  Arms: Night shift protocol with diet A; Night shift protocol with diet B

SUMMARY:
The goal of this clinical trial is to test whether food timing impacts metabolic health in healthy participants.

Participants will:

* complete 2 inpatient stays
* be provided with test meals
* have frequent blood draws

DETAILED DESCRIPTION:
The investigators aim to investigate the influence of different food timing, without changing 24-h caloric and nutrient intake, on glucose and fat tolerance and energy expenditure in healthy people on a simulated day or night shift.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no acute or chronic medical and psychiatric disorders
* BMI: 18.5-29.9 kg/m2

Exclusion Criteria:

* Smokers, current tobacco or e-cigarette use
* Drug or alcohol dependency
* Pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in glucose tolerance between Meal Conditions and Shift Work | 24 hours
  Glucose incremental area under the curve (AUC) from mixed meal tests
Difference in diet-induced thermogenesis between Meal Conditions and Shift Work | 24 hours
  Postprandial energy expenditure incremental area under the curve (AUC) from mixed meal tests
Difference in plasma triglyceride level between Meal Conditions and Shift Work | 24 hours
  Triglyceride area under the curve (AUC) over 24 hours

SECONDARY OUTCOMES:
Difference in insulin sensitivity between Meal Conditions and Shift Work | 24 hours
  Insulin sensitivity index derived from Oral Minimal Model
Difference in beta-cell function between Meal Conditions and Shift Work | 24 hours
  Beta-cell function index derived from Oral Minimal Model
Difference in 24-h glycemia between Meal Conditions and Shift Work | 24 hours
  Glucose area under the curve (AUC) based on CGM over 24 hours
Difference in postprandial incretin level between Meal Conditions and Shift Work | 24 hours
  Incretin incremental area under the curve (AUC) from mixed meal tests
Difference in substrate oxidation between Meal Conditions and Shift Work | 24 hours
  Postprandial substrate oxidation incremental area under the curve (AUC) from mixed meal tests
Difference in plasma free fatty acids level between Meal Conditions and Shift Work | 24 hours
  Free fatty acids area under the curve (AUC) over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Frank Scheer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No